CLINICAL TRIAL: NCT06403618
Title: Evaluation of the PreCursor-M+® Assay Performance in the Management of Women Diagnosed With CIN2
Brief Title: Evaluation of the PreCursor-M+® in CIN2
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4438
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collection of liquid based cervical samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- active surveillance: wait-and-see strategy
- immediate treatment: surgical treatment per clinical practice

SUMMARY:
The goal of this observational study is to to evaluate the accuracy and sensitivity of PreCursor-M+ on a post-aliquot of liquid-based cytology (LBC) cervical samples (biopsy) obtained by physicians in a group of women with histologically-proven diagnoses of CIN2.

The PreCursor-M+® assay is a multiplex real-time methylation specific PCR test that identifies the level of promotor methylation of the host cell genes FAM19A4 and miR124-2, known biomarkers associated with cervical carcinoma and transforming CIN in cervical cells.

To evaluate the clinical course of CIN2 at 2 years after the first diagnosis, with an interval evaluation at 6 months.

After enrolment, women will be divided into two groups: "active surveillance" and "immediate treatment". In the first group, clinical outcomes to be assessed, in relation to the PreCursor-M+ result at baseline, will include regression to <CIN2, persistence of CIN2, and progression to CIN3+. In the second group, we will evaluate the histological diagnosis at cone specimen (downgrading or upgrading) and the 2-year cumulative incidence of CIN2+ recurrence based on the PreCursor-M+ result at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. age at diagnosis of 18 years or older;
2. histological confirmation of CIN2 after colposcopic-guided cervical biopsy or conservative surgical treatment, including loop electrosurgical excision procedure (LEEP) and laser conization;
3. known HPV test result at baseline;
4. ability to understand and sign the informed consent;
5. written informed consent given.

Exclusion criteria:

1. unknown HPV test result at diagnosis;
2. vulnerable patients.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: women with histological diagnosis of CIN2
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2027-06-17 (Estimated)

PRIMARY OUTCOMES:
Evaluation of methylation of the host cell genes FAM19A4 and miR124-2 | 6 months
  The PreCursor-M+® assay is a multiplex real-time methylation specific PCR test that identifies the level of promotor methylation of the host cell genes FAM19A4 and miR124-2, known biomarkers associated with cervical carcinoma and transforming CIN in cervical cells. This test can identify patients with spontaneous regressing precancer lesions (negative result) from patients with a progressing precancer lesion (positive result).

SECONDARY OUTCOMES:
Evaluation of clinical course of CIN2 at 2 years after diagnosis | 2 years
  To evaluate the clinical course of CIN2 at 2 years after the first diagnosis, with an interval evaluation at 6 months. After enrolment, women will be divided into two groups: "active surveillance" and "immediate treatment". In the first group, clinical outcomes to be assessed, in relation to the PreCursor-M+ result at baseline, will include regression to <CIN2, persistence of CIN2, and progression to CIN3+. In the second group, we will evaluate the histological diagnosis at cone specimen (downgrading or upgrading) and the 2-year cumulative incidence of CIN2+ recurrence based on the PreCursor-M+ result at baseline.
Evaluation of overall accuracy of PreCursor-M+ | 6 months - 2 years
  Overall accuracy, positive predictive value and negative predictive value of PreCursor-M+

CONTACTS AND LOCATIONS:
Overall Officials: Anna Daniela Iacobone, Principal Investigator — European Institute of Oncology
Locations (2):
- Italy (2):
  - European Institute of Oncology, Milan,, Milan
  - European Institute of Oncology, Milan